CLINICAL TRIAL: NCT07346144
Title: A Phase I/II Study of an AAV-1 Mediated Dual-Payload Gene Therapy in Patients With High Grade Glioma
Brief Title: Study of an AAV Mediated Dual-Payload Gene Therapy in Patients With High Grade Glioma
Acronym: ADePT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Trogenix ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TGX-CS-701
Record Dates: First submitted 2026-01-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma (GBM); High Grade Gliomas; Recurrent Glioblastoma; Newly Diagnosed Glioblastoma
Keywords: Glioblastoma; Immunotherapy; Gene Therapy; AAV; HSV-tk; IL-12; TGX-007
MeSH Terms: conditions — Glioblastoma | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Finding (Experimental): Dose escalation (with dose levels -1, 1, 2)
  Interventions: Drug: TGX-007; Drug: Valaciclovir
- Newly Diagnosed Expansion (Experimental): Expansion in Newly Diagnosed High Grade Glioma patients at the Optimal Biological Dose.
  Interventions: Drug: TGX-007; Drug: Valaciclovir
- Recurrent Glioblastoma Expansion (Experimental): Expansion in recurrent glioblastoma patients at the Optimal Biological Dose.
  Interventions: Drug: TGX-007; Drug: Valaciclovir

INTERVENTIONS:
Drug: TGX-007 — TGX-007 administered as single intratumoural injection
Drug: Valaciclovir — Oral valaciclovir administered 3 times daily for 14 - 21 days

SUMMARY:
The goal of this clinical trial is to first define the Safety and Optimal Biological Dose (OBD) of study drug TGX-007 and to then further investigate the safety and efficacy in patients with newly diagnosed or recurrent Glioblastoma.

TGX-007 is a gene therapy drug delivered by a harmless adeno-associated virus (AAV) vector which delivers two combined therapeutic payloads to enable killing of proliferative cells and activation of an anti-tumour immune response. One is herpes simplex virus thymidine kinase (HSV-tk), which converts the pro-drug valaciclovir into an active drug that can kill tumour cells and the other is interleukin 12 (IL-12), which activates the body's immune system to recognise and fight the tumour.

Patients newly diagnosed with glioblastoma suitable for standard of care surgery and chemoradiotherapy or patients with recurrent glioblastoma suitable for further surgery may be eligible for the study. Patients will receive TGX-007 by a direct intratumoural injection and will then take the pro-drug valacyclovir orally for up to 21 days before proceeding to standard of care surgery.

The study is split into two phases. Phase I will treat patients at different dose levels of TGX-007 to identify the Optimal Biological Dose that will be used to further expand the study into Phase II. Phase II will expand the number of patients treated at the selected OBD to investigate how effective TGX-007 is at treating newly diagnosed and recurrent GBM.

Approximately 68 people aged 18-70 will take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years
* Karnofsky performance status ≥70
* Newly diagnosed patients: Unifocal, unilateral high-grade glioma based on MRI
* Recurrent patients: First radiological progression (as determined by the multidisciplinary team [MDT]) of GBM previously treated with standard care surgery and chemoradiotherapy. Patients must have a prior confirmed histological/molecular diagnosis of GBM
* Newly diagnosed patient: suitable for six weeks of chemoradiotherapy followed by six months of adjuvant temozolomide (Stupp protocol)
* Debulking surgery is indicated for optimal patient care
* Able to swallow oral medication
* Willing to avoid live vaccines
* Adequate organ function
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to Day 0.
* All patients must agree to practice true abstinence or to use highly effective contraception
* Patient is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Patient who is pregnant, lactating or planning pregnancy during the course of the study
* Immunodeficiency or active auto-immune disease requiring systemic therapy.
* Active viral, bacterial or fungal infection requiring concurrent antivirals or antibiotics within 7 days of surgery
* Live vaccine within 28 days prior to Day 0
* Use of immunosuppressant or immune modulatory medicines within 28 days prior to Day 0
* History of tuberculosis infection or chest x-ray or computed tomography (CT) chest showing radiological evidence of previous tuberculosis infection
* Received previous treatment with a gene therapy
* Significant history of a central nervous system disorder that, in the opinion of the Investigator, would preclude enrolment
* Major surgery within 28 days prior to Day 0. A stereotactic biopsy is permitted
* Known hypersensitivity or contraindications to valaciclovir, gadolinium, or any excipients for TGX-007
* Contraindication to MRI with gadolinium
* Any condition expected to interfere with the intended timing of debulking surgery
* Previous non-glioma cancer within 3 years (other than treated squamous/basal cell skin cancer, treated early-stage cervical cancer or treated/biochemically stable, organ confined prostate cancer)
* Any other significant disease or disorder which, in the opinion of the Investigator, may put the patient at risk because of participation in the study or may influence the results of the study or the patient's ability to participate in the study
* Patients who have participated in another research study involving an investigational product in the past 12 weeks or 5 half-lives of the product
* Any psychological, familial, sociological, or geographical consideration potentially hampering compliance with the study protocol and follow up schedule; these conditions should be discussed with the patient before registration in the study
* Unwilling to allow their general practitioner, if appropriate, to be notified of participation in the study

Newly diagnosed patients only:

* Any prior therapy for glioma
* Intended use of tumour treating fields

Recurrent patients only:

* Prior toxicities from anti-cancer agents or radiotherapy which have not recovered to ≤Grade 1 severity
* Intended use of tumour treating fields

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of TGX-007 when administered to patients with newly diagnosed HGG or recurrent GBM and to identify the OBD | Day 0 (TGX-007 injection) to 28 days post administration of TGX-007
  Incidence of AEs/SAEs, incidence of DLT within 28 days of TGX-007 administration at each dose level, and incidence of HSV-tk mRNA expression, or equivalent, in tissue
Overall Survival rate of patients with newly diagnosed HGG or recurrent GBM treated with TGX-007 | Day 0 (TGX-007 injection) to 18 months (newly diagnosed); Day 0 (TGX-007 injection) to 6 months (recurrent patients)
  Overall Survival at 18 months (newly diagnosed patients) and 6 months (recurrent patients).

SECONDARY OUTCOMES:
Overall Survival | Baseline to 5 year follow up
  Median OS and OS up to 5 years by Kaplan-Meier analysis.
Viral shedding in body fluids following delivery of TGX-007. | Baseline until 3 consecutive negative samples, assessed up to 5 years post treatment.
  Detection of vector genomes by droplet digital polymerase chain reaction (ddPCR) in patient samples
Progression-free survival (PFS) of patients with newly diagnosed HGG or recurrent GBM treated with TGX-007. | Date of surgery to the earliest date progression is documented or death from any cause, measured out to 5 years post surgery
  PFS as determined by the Investigator
Objective response rate (ORR) of patients with newly diagnosed HGG or recurrent GBM treated with TGX-007. | Baseline to 21 days
  ORR on pre-operative MRI per Response Assessment in Neuro-Oncology 2.0 (RANO 2.0) criteria.
Assess the safety and tolerability of TGX-007 when administered to patients with newly diagnosed HGG or recurrent GBM | Baseline to 5 year follow up
  Incidence of AEs/SAEs.

CONTACTS AND LOCATIONS:
Locations (2):
- Ohio State University Hospital, Columbus, Ohio, United States
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No